CLINICAL TRIAL: NCT03951558
Title: Comparison of the Impact of Nutritional Treatment vs Hydrochlorothiazide on Bone Mineral Density and Body Composition in Children With Idiopathic Hypercalciuria of the Hospital Infantil de Méxio Federico Gómez
Brief Title: Comparison of the Impact of Diet vs Thiazide in BMD in Children With Idiopathic Hypercalciuria
Acronym: HIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Mara Medeiros, Ph D Mara Medeiros Domingo, Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HIM-2017-046
Record Dates: First submitted 2019-05-10; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Hypercalciuria; Idiopathic; Nephrolithiasis
Keywords: diet; drinking water; salt; dietaryprotein
MeSH Terms: conditions — Hypercalciuria; Nephrolithiasis | interventions — Diet; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant
Masking Description: The capsules are the same color in the placebo group and the intervention group. The content of the capsules is similar in both groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diet for calciuria prevention (Experimental): placebo capsules and a strict eating plan will be given. The placebo will look similar to that of hydrochlorothiazide and will be prepared in the Nephrology Research Laboratory by Biol. Ana María Hernández Sánchez and Quim Lourdes Ortiz.
  Interventions: Other: Diet for calciuria prevention
- hydrochlorothiazide for calciuria prevention (Placebo Comparator): recommendations for water intake and decrease in salt intake will be given.
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Other: Diet for calciuria prevention — Dietary recommendations for water, salt, calcium and proteins according to age and DIR
  Other Names: Diet for hypercalciuria
  Arms: Diet for calciuria prevention
Drug: Hydrochlorothiazide — Hydroclorothiazide recommendations for hypercalciuria
  Other Names: Hydroclorothiazide in hypercalciuria
  Arms: hydrochlorothiazide for calciuria prevention

SUMMARY:
The investigator's objective is to compare and evaluate the impact of nutritional treatment vs. pharmacological treatment (hydrochlorothiazide) in bone mineral density in children with idiopathic hypercalciuria.

A randomized, open-label, one-year follow-up study will be conducted in children aged 5 to 21 years with a confirmed diagnosis of idiopathic hypercalciuria or lithiasis, excluding those patients with secondary hypercalciuria (primary hyperoxaluria, treatment with vitamin D, Bartter syndrome, primary hyperparathyroidism), previous kidney transplantation. The impact of diet (hyposodic, calcium intake according to DIR for age, normal protein intake and high water intake) will be evaluated vs. the pharmacological treatment (hydrochlorothiazide) on bone mineral density.

DETAILED DESCRIPTION:
A randomized, open-label clinical trial will be conducted with a one-year follow-up. For which basal measurement of calciuria, citraturia, serum creatinine, serum and urinary electrolytes, parathyroid hormone, vitamin D levels and renal ultrasound, as well as dietary intake (protein, energy, salt and water). The dietary intake per day of food and pharmacological treatment will be evaluated quarterly, body composition (anthropometry) and serum and urinary electrolyte levels will be measured; Bone constitution (DXA, quantitative bone ultrasound), IL-1 (as inflammatory markers) and vitamin D will be evaluated every six months.

Participants will be blinded to the pharmacological treatment they will receive. The randomization of the participants will be done through the page www.randomization.com. The randomization was performed by blocks, where blocks of 6 members each were made i. Group 1: only recommendations of water intake and reduction of salt intake and hydrochlorothiazide will be given (the dose will be assigned according to weight and sex by a pediatric nephrologist, dose of 0.5-1.5mg / kg / day, starting with the dose 1 mg / kg). Hydrochlorothiazide will be provided to the patient.

ii. Group 2: placebo capsules and a strict diet plan will be given. The placebo will look similar to that of hydrochlorothiazide and will be prepared in the Nephrology Research Laboratory by Biol. Ana María Hernández Sánchez and Quim Lourdes Ortiz. The feeding plan will be appropriate for the patient, it will consist of:

1. 40 ml / Kg / day of water
2. Protein according to age and sex
3. Recommendations for low sodium intake
4. Calcium according to age and sex (minimum 800mg)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic hypercalciuria
* Man or women
* 5 to 21 years

Exclusion Criteria:

* Clinical diagnosis of secondary hypercalciuria (primary hyperoxaluria, treatment with vitamin D, Bartter syndrome, primary hyperparathyroidism)
* Previous kidney transplant
* Clinical diagnosis of kidney disease.
* Vitamin D intake (more than 800 mg/day)

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-05-11 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
bone mineral density | one year
  bone mineral density will be evaluated by means of score z evaluated by dexa

SECONDARY OUTCOMES:
Ca/Cr index | one year
  urinary calcium excretion will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ortiz, Master, Study Chair — Laboratorio de Enseñanza Virtual y Ciberpsicología. Facultad de Psicología. UNAM
Locations (1):
- Children's Hospital of Mexico, Federico Gómez, México, México City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
a report of results will be made by means of a research article and information will be provided that researchers interested in the obtained data request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: will be available at within one year
Access Criteria: Requests for additional information will be reviewed by Nutriologa Ma Elena Ortiz and PhD. Mara Medeiros Domingo